CLINICAL TRIAL: NCT02417701
Title: A Phase 2 Study of MLN0128 (TAK-228) in Patients With Advanced Non-Small Cell Lung Cancers Harboring NFE2L2 and KEAP1 Mutations
Brief Title: Sapanisertib in Treating Patients With Stage IV or Recurrent Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00545; NCI-2015-00545 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-249; 2015-00500; 9780 (Other: Memorial Sloan Kettering Cancer Center); 9780 (Other: CTEP); P30CA008748 (NIH)
Record Dates: First submitted 2015-04-14; First posted 2015-04-16 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Lung Squamous Cell Carcinoma; Stage IV Lung Squamous Cell Carcinoma AJCC v7
MeSH Terms: interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sapanisertib) (Experimental): Patients receive sapanisertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sapanisertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228

SUMMARY:
This phase II trial studies how well sapanisertib works in treating patients with lung cancer that is stage IV or has come back (recurrent) and has a mutation in the NFE2L2, KEAP-1, or KRAS gene. Damage to these genes may cause the cancer to grow. Sapanisertib may stop this from happening by blocking enzymes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the overall response rate of the TORC1/TORC2 inhibitor sapanisertib (MLN0128 [TAK-228]) in stage IV squamous cell lung cancers or KRAS mutant lung cancers harboring NFE2L2 or KEAP1 mutations.

SECONDARY OBJECTIVES:

I. To evaluate the median progression free survival of patients in each cohort. II. To explore the feasibility of performing reverse phase protein array analysis (RPPA) in paired snap-frozen core biopsies from patients in this study prior to MLN0128 (TAK-228) dosing and during week 2 of treatment.

III. To describe the effectiveness of MLN0128 (TAK-228) in suppressing activation of mTOR and PI3K signaling through the exploratory RPPA analysis.

OUTLINE:

Patients receive sapanisertib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV or recurrent squamous cell lung cancer or KRAS mutant lung cancer that harbors any of the NFE2L2 mutations or KEAP1 mutations; any KEAP1 mutation will be eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have completed at least 1 prior line of systemic therapy; patients who have declined first line therapy or for whom first-line therapy would be clinically inappropriate, will be considered eligible for the trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Fasting serum glucose =< 130 mg/dL or hemoglobin A1C (HBA1C) < 7.0%
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients with controlled diabetes are allowed on study; controlled diabetes is defined as fetal bovine serum (FBS) =< 130 mg/dL in the context of this study
* The effects of MLN0128 (TAK-228) on the developing human fetus are unknown; for this reason women of child-bearing potential and men must agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method, at the same time, prior to study through 90 days (or longer, as mandated by local labeling [e.g., United States Package Insert (USPI), Summary of Product Characteristics (SmPC), etc;]) after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; any woman who becomes pregnant while receiving MLN0128 (TAK-228) will be removed from the trial; men treated or enrolled on this protocol must also agree to use highly effective barrier contraception prior to the study, for the duration of study participation, and 120 days after completion of MLN0128 (TAK-228) administration; men must agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow oral medications
* Known human immunodeficiency virus (HIV) positive patients who meet the following criteria will be considered eligible:

  * CD4 count > 350 cells/mm^3
  * Undetectable viral load
  * Maintained on modern therapeutic regimens utilizing non-CYP-interactive agents

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to the planned start of study treatment or those who have not recovered to baseline or less than grade 2 from adverse events from prior treatments
* Patients who are receiving any other investigational agents
* Patients with untreated central nervous system (CNS) metastases; patients with treated CNS metastases who are off steroids are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN0128 (TAK-228)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; no ischemic myocardial or cerebrovascular event, class III or IV heart failure, placement of pacemaker, or pulmonary embolism within six months of receiving first dose of MLN0128 (TAK-228)
* Baseline prolongation of the rate-corrected QT interval (QTc) > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes
* Pregnant women are excluded from this study because MLN0128 (TAK-228) is an mTOR agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MLN0128 (TAK-228), breastfeeding should be discontinued if the mother is treated with MLN0128 (TAK-228)
* Patients previously treated with an mammalian TOR (mTOR) or PI3K inhibitor
* Concomitant administration of any proton pump inhibitor (PPI) is not permitted during the study; patients receiving PPI therapy before enrollment must stop using the PPI for 7 days before their first dose of study drugs
* Uncontrolled diabetes mellitus (fasting plasma glucose > 130 mg/dL despite optimal medical management of hyperglycemia)
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
* Patients receiving histamine H2 receptor antagonists before enrollment must stop using these medications for at least 24 hours before their first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Paik, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sapanisertib)
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 68.52 [46 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Response [CR] + Partial Response [PR])
Description: Overall response rate (CR+PR) will be calculated separately for each cohort, including exact 95% confidence intervals. Duration of overall response and duration of stable disease will be calculated and summarized. Overall response rate was determined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1). Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: CT imaging was obtained after every 2 cycles, or 8 weeks, starting from cycle 1 day 1 until end of study treatment, up to 1 year.
Population: The number of participants analyzed for ORR is the response evaluable cohort as defined by the protocol, which is a subset of the total study population reflected in the participant flow module.
Measure: Count of Participants; unit: Participants
Groups:
- NFEL2 Squamous Cohort; KEAP1 Squamous Cohort; KRAS/NFE2L2 or KEAP1 NSCLC Cohort: Patients receive sapanisertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | NFEL2 Squamous Cohort | KEAP1 Squamous Cohort | KRAS/NFE2L2 or KEAP1 NSCLC Cohort
Number analyzed (Participants) | 12 | 6 | 6
Participants
  ORR: Complete Response + Partial Response | 3 | 1 | 0
  No ORR | 9 | 5 | 6

2. Secondary Outcome: Progression-free Survival
Description: Median progression-free survival will be estimated using the Kaplan-Meier method with a two-sided 95% confidence interval. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a unequivocal increase in a non-target lesion, or the appearance of new lesions
Time Frame: From start of treatment (cycle 1 day 1) until the date of first documented progression or death, over the trial enrollment period, up to 1 year.
Population: PFS in the secondary outcome section is the response evaluable cohort, which is a subset of the total study population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NFEL2 Squamous Cohort | KEAP1 Squamous Cohort | KRAS/NFE2L2 or KEAP1 NSCLC Cohort
Number analyzed (Participants) | 12 | 6 | 6
months | 8.9 [5.6 to NA] — Upper limit was not reached due to insufficient number of participants with events | 3.7 [1.8 to NA] — Upper limit was not reached due to insufficient number of participants with events | 2.1 [1.6 to NA] — Upper limit was not reached due to insufficient number of participants with events

3. Secondary Outcome: Feasibility of Reverse Phase Protein Array Analysis, Defined as the Ability to Procure Sufficient Quantity and Quality of Tumor Protein for Sample
Description: Single target signaling changes will be reported as percentages relative to the baseline pre-treatment tumor sample. Larger scale pathway changes will qualitatively represented through heatmaps.
Time Frame: Up to week 2
Population: Data were not collected
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Treatment (Sapanisertib)
All-Cause Mortality (participants affected / at risk) | 6/34
Serious Adverse Events (participants affected / at risk) | 8/34
Other Adverse Events (participants affected / at risk) | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sapanisertib) (N=34)
Diarrhea (Gastrointestinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Thromboembolic event (Vascular disorders) | 3
Creatinine Increased (Investigations) | 2
Mucositis (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sapanisertib) (N=34)
Hyperglycemia (Metabolism and nutrition disorders) | 21
Fatigue (General disorders) | 11
Diarrhea (Gastrointestinal disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Weight loss (Investigations) | 8
Mucositis oral (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5
Platelet count decreased (Investigations) | 5
Cholesterol high (Investigations) | 3
Flatulence (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02417701/Prot_SAP_000.pdf